CLINICAL TRIAL: NCT05015036
Title: Evaluation of an Enhanced Recovery Protocol After Minimally Invasive Lumbar Surgery.
Acronym: ERAMIS
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02669-30
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Spine Surgery
MeSH Terms: interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive surgery of the lumbar spine with ERAS: Minimally invasive surgery of the lumbar spine with Enhanced Recovery After Surgery (ERAS)
  Interventions: Procedure: ERAS
- Minimally invasive surgery of the lumbar spine: Minimally invasive surgery of the lumbar spine
  Interventions: Procedure: Minimally invasive surgery

INTERVENTIONS:
Procedure: ERAS — Minimally invasive surgery of the lumbar spine with Enhanced Recovery After Surgery (ERAS)
  Groups: Minimally invasive surgery of the lumbar spine with ERAS
Procedure: Minimally invasive surgery — Classic Minimally invasive surgery of the lumbar spine
  Groups: Minimally invasive surgery of the lumbar spine

SUMMARY:
Prospective longitudinal multicentre observational study carried out on a population of patients undergoing minimally invasive spine surgery and divided into two parallel cohorts according to the presence or absence of a Enhanced Recovery After Surgery (ERAS) programme.

The patient will be assessed during 4 visits: At inclusion before surgery, at D0 (day of surgery), at D1 (postoperative visit) and at M1 (follow-up visit).

DETAILED DESCRIPTION:
On a population of patients undergoing minimally invasive lumbar spine surgery divided into two cohorts of equal size according to the presence or absence of a Enhanced Recovery After Surgery (ERAS) programme:

Primary objective To compare the percentage of therapeutic success achieved in each group one month after surgery.

Secondary objectives: to compare between groups:

* Postoperative pain intensity at D1 and M1
* Analgesic consumption (in stages) at D1 and M1
* Pain-free walking distance at M1
* Surgery conditions (duration of operation, duration of hospitalisation)
* Frequency of adverse events related to surgery (infection rate, 1 month recovery rate, transfusion requirements)
* Emotional impact of the management

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (18 years or older)
* Patient who has agreed to participate in the study and has read and signed the consent form for participation in the study
* Patient for whom a minimally invasive spine surgery is planned: (dicectomy, lumbar canal recalibration with or without laminectomy, lumbar arthrodesis by posterior approach limited to one stage)

Exclusion Criteria:

* Patient with a contraindication to spinal anaesthesia
* A bedridden or institutionalised patient
* Mental deficiency or any other reason that may hinder the understanding or the strict application of the protocol
* Patient not affiliated to the French social security system
* Patient under legal protection, guardianship or curatorship
* Patient already included in another therapeutic study protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient population for minimally invasive lumbar spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index improvement | Month 1
  The Oswestry Disability Index (Appendix 1) (also known as the Oswestry Low Back Pain Disability) is the gold standard tool for assessing functional disability related to low back pain and functional recovery after surgery. It consists of ten questions rated from 0 to 5 (from most to least favourable). The result is expressed as a percentage according to the following formula [score obtained / (maximum score)] X 100. The maximum score is 50 if all the questions have been filled in, 45 if one question has not been filled in etc..... The disability rate, corresponding to the percentage, obtained is considered minimal between 0 and 20%, moderate between 21 and 40% and severe above 41%.
  Therapeutic success defined as an improvement ≥30% in the Oswestry Disability Index between initial and final visit is the primary endpoint

SECONDARY OUTCOMES:
Post-operative pain | Day 1
  The intensity of the pain will be assessed using a simple numerical scale (ENS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Post-operative pain | Month 1
  The intensity of the pain will be assessed using a simple numerical scale (ENS) graduated from 0 (no pain) to 10 (worst pain imaginable).
Consumption of level I, II and II analgesics | Day 1
  Consumption of level I, II and II analgesics. Count of treatments
Consumption of level I, II and II analgesics | Month 1
  Consumption of level I, II and II analgesics
Pain-free walking perimeter | Month 1
  Measurement in meters of the distance the patient travels until he/she is forced to stop due to pain
Evolution of Hospital Anxiety and Depression (HAD) scale score and sub-scores | Month 1
  The emotional impact of the disease will be more precisely evaluated by the Hospital Anxiety and Depression (HAD) questionnaire, a screening tool for the most common manifestations of anxiety and depressive disorders to be completed by the patient. The scale comprises 14 questions, with 7 items assessing anxiety and 7 items assessing depression.
  A minimum score of 10 on one of the sub-scores was retained as a criterion for detecting depressive or anxious manifestations. The HAD questionnaire will be completed by the patient at the inclusion visit (V1) and at the end of the study (V4).
Duration of intervention | Day 1
  Duration of the surgery in hours
Length of hospital stay | Month 1
  Length of hospital stay in days
Adverse events related to surgery | Month 1
  All adverse events related to surgery will be collected and compared in the 2 groups
Visual Analogue Scale overall patient satisfaction | Month 1
  The patient's satisfaction with his or her treatment and results will be assessed at the end of the study on a visual analogue scale graduated from 0 (very dissatisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur ANDRE, MD, Principal Investigator — Clinique Geoffroy Saint-Hilaire
Locations (1):
- Clinique Geoffroy Saint-Hilaire, Paris, France

IPD SHARING:
Plan to Share IPD: No